CLINICAL TRIAL: NCT05521334
Title: Clinical Evaluation of MicroPulse Transscleral Laser Cyclophotocoagulation With the Zig Zag Mode of Application in Adult Glaucomatous Patients
Brief Title: MicroPulse Transscleral Laser Cyclophotocoagulation With the Zig Zag Mode in Glaucoma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Ahmed Samy Abohussein, principal investigator, Helwan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahmed Sami Ahmed
Record Dates: First submitted 2022-08-03; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Refractory Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Adult Glaucomatous patients with refractory glaucoma (Experimental): Adult glaucomatous patients with uncontrolled intraocular pressure despite maximal tolerated medical treatment
  Interventions: Device: micropulse transscleral cyclophotocoagulation

INTERVENTIONS:
Device: micropulse transscleral cyclophotocoagulation — glaucomatous patients with uncontrolled intraocular pressure (despite maximal tolerated anti-glaucoma medical treatment) were selected for micro-pulse trans-scleral cyclophotocoagulation using an MP3 handpiece with Iridex Cyclo G6 Laser settings (2000mW of 810 nm infrared diode laser set on micro-pulse delivery mode with 31.3 % duty cycle). The laser will be delivered over three quadrants for 90 seconds for each quadrant (total 270 sec) in Zigzag mode sparing the fourth quadrant for either further intervention or a previous surgery performed. Follow up examination (for at least 6 months) will include assessment of IOP in terms of percentage of IOP reduction and sustainability of results, BCVA, and the number of medications post-operatively.

SUMMARY:
This is a prospective single-arm clinical trial in which patients with neovascular or primary open angle glaucoma with uncontrolled intraocular pressure (despite maximal tolerated anti-glaucoma medical treatment) were selected for micro-pulse trans-scleral cyclophotocoagulation using an MP3 handpiece with Iridex Cyclo G6 Laser settings (2000mW of 810 nm infrared diode laser set on micro-pulse delivery mode with 31.3 % duty cycle). The laser will be delivered over three quadrants for 90 seconds for each quadrant (total 270 sec) in Zigzag mode sparing the fourth quadrant for either further intervention or a previous surgery performed. Follow up examination (for at least 6 months) will include assessment of IOP in terms of percentage of IOP reduction and sustainability of results, BCVA, and the number of medications post-operatively.

DETAILED DESCRIPTION:
From the expert opinion, using the ZigZag technique would increase the success rate by 10-20 %.

Type of study: Prospective single arm clinical trial. Participants: 24 eyes of 20 consecutive patients who underwent MP-TSCPC with Zig Zag technique at a private ophthalmology center from March 16,2021 to April 12,2021 and who had at least 6 months of follow-up were included.

All cases were performed in a specialized ophthalmic center in Cairo, Egypt by the same surgeon with the same technique and standardized parameters.

On presentation, proper history was taken from all patients including personal history, history of systemic illness, family history for glaucoma, past ocular history, history of current illness including onset, course, duration of disease, causes of progression and current medication.

Ophthalmic examinations included best corrected visual acuity, anterior segment, posterior segment, gonioscopy and measuring intraocular pressure.

Investigations performed included visual fields which although being important for diagnosis, they could not be done in the majority of cases as VA was severely affected as will be clarified in the results section, OCT optic nerve head, and measurement of central corneal thickness in addition to ocular ultrasonography if fundus could not be examined to detect the pathology and document the retinal condition.

All the data were documented to be compared to post-operative results as IOP reduction, complications and number of medications.

Surgical procedure:

All surgeries were done under peri-bulbar blockage with short duration anesthetic (2% lidocaine) with systemic sedation for ocular anesthesia and akinesia.

Lubricant gel was used to facilitate probe motion.

Micro-pulse TSCPC was done using an MP3 handpiece (IRIDEX, CYCLO G6 Glaucoma Laser System, Mountain View, CA) with Laser settings (2000-mW of 810-nm infrared diode laser set on micro-pulse delivery mode with 31.3 % duty cycle where on-cycle of 0.5-ms followed by off-cycle of 1-ms).

The laser was delivered in Zigzag pattern respecting the anatomy of cilliary body being 6mm in length, and the probe is formulated thus the fiber optic is projected for 0.7 mm with contact diameter of 600 µ placed 3 mm from the limbus, the idea is to cover the largest diameter of ciliary body and ciliary processes putting into consideration the normal variation in ciliary body length and position, so the probe is moved for 2 mm perpendicular to a line 3 mm circumferential to the limbus so as to cover the largest circumference of the area supposed to hinder the cilliary body over three quadrants for 90 seconds for each quadrant (total 270 sec) sparing the fourth quadrant for either further intervention or a previous surgery performed (in all cases the 2 inferior quadrants were treated in addition to superotemporal quadrant being more accessible for Zig Zag pattern sparing the superonasal quadrant for further inrtervention except if a previous glaucoma surgery was performed in supertemporal quadrant where the superonasal quadrant was treated).]

Follow up examination (for at least 6 months) included assessment of IOP in terms of percentage of IOP reduction and sustainability of results, BCVA, the number of medications post-operatively, and reported complications.

Success was defined as either maintaining an IOP of less than 21 mmHg or achieving a reduction of 30% from baseline IOP with or without supplementing topical anti-glaucoma medications which was further classified as complete success where criteria of success were achieved without the need to add antiglaucoma medications, and qualified success where the antiglaucoma medications were needed to reach the target IOP

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with uncontrolled intraocular pressure
* on maximally tolerated medical treatment.
* Primary open angle glaucoma or neovascular glaucoma

Exclusion Criteria:

* patients with other types of glaucoma.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Measuring the of intraocular pressure (in mmHg) using Goldman applanation tonometer to calculate the percentage of reduction. | 6 months
  Intraocular pressure will be measured in (mmHg) using Goldman applanation tonometer (an instrument that is based on Imbert-Fick law. It is considered to be the gold standard instrument for measurement of Intraocular pressure (IOP).It was named after Austrian-Swiss ophthalmologist Hans Goldmann ) before the procedure then measured in the 1 week follow up , 1 month , 3 months and 6 months follow up where each measure will be divided by the preoperative IOP to calculate the percentage of intra ocular pressure reduction and monitor the stability of IOP.
  the success rate will be calculated depending on the rate of IOP reduction in the last follow up.

CONTACTS AND LOCATIONS:
Overall Officials: TareK Aboulnasr, MD, Study Director — Benha University
Locations (1):
- Helwan University, Helwan, Egypt